CLINICAL TRIAL: NCT07289867
Title: Nutritional Effects of Supplementing Nonagenarians With a Supplement Based on a Fruit From the Cerrado: Buriti
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Sergio Henrique Sousa Santos, Professor / principal investigator, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 6.790.431
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Malnutrition in the Elderly
Keywords: Nonagenarians; malnutrition; Cerrado; nutritional supplements
MeSH Terms: conditions — Malnutrition | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This randomized clinical trial included 40 eligible participants, randomly assigned into two groups of 20. One group received a buriti-based supplement (Supplement Test - ST), while the control group received capsules containing the same vitamins and minerals (Vitamin Mix - VM). The intervention lasted 12 weeks, during which participants were evaluated before and after for nutritional status using the HAND test, anthropometric measurements, handgrip strength (HGS), and biochemical blood tests.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement Group (Experimental): Participants received the supplement test (Nutricer Energia Zero-lactose) daily for 3 months
  Interventions: Dietary Supplement: Nutricer Energia Zero-lactose
- Control Group (Multivitamin Mix) (Active Comparator): Participants received a multivitamin mix daily for 3 months
  Interventions: Dietary Supplement: Multivitamin Mix

INTERVENTIONS:
Dietary Supplement: Nutricer Energia Zero-lactose — Daily administration of two tablespoons of solubilized in whole milk once a day for 3 months.
  Other Names: Supplement Group
  Arms: Supplement Group
Dietary Supplement: Multivitamin Mix — Daily administration of one multivitamin capsule for 3 months.
  Other Names: Control Group (Multivitamin Mix)
  Arms: Control Group (Multivitamin Mix)

SUMMARY:
The population aged over 90 is growing worldwide, and the search for strategies to promote a better quality of life for the older persons is a challenge for science. Advancing age is associated with several physiological changes leading to different diseases, among which malnutrition and sarcopenia stand out. Malnutrition prevention and treatment are based on functional food/nutritional interventions, such as oral supplement use. However, studies evaluating the effectiveness of these supplements in nonagenarians are still scarce in the literature. The present study aimed to evaluate the use of a buriti fruit (Mauritia flexuosa) supplement in persons 90 years and older. The study included 40 individuals who were randomized into two groups. The group Supplement Test (ST) used a Buriti-based supplement with full vitamins and minerals; the control group used a capsule containing the same composition of vitamins and minerals as the test supplement, which was called Vitamin Mix (VM). The intervention lasted 12 weeks. The following analyses were carried out before and after this period: Mini Nutritional Assessment (MNA) questionnaire, handgrip strength (HGS), biochemical tests, and anthropometric measurements. The main results showed that the Buriti supplement led to a significant increase in body weight, Body Mass Index (BMI), handgrip strength, and globulins, when compared to the group that used the vitamin mix. Therefore, it can be concluded that the buriti supplement promotes an improvement in body composition, increased strength, and globulins in nonagenarians, and may be a viable and effective strategy for malnutrition treatment.

ELIGIBILITY:
Inclusion Criteria:

Participants aged 90 or over were selected from the database of the Reference Center for Elderly Health Care in Montes Claros, MG .

Exclusion Criteria:

* Exclusion criteria included severe obesity, decompensated chronic diseases, or inability/refusal to consent.

Min Age: 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Body Weight | Baseline and after 12 weeks of supplementation
  Body weight (kg) was measured using a calibrated digital scale to evaluate changes after supplementation.
Change in Muscle Strength | Baseline and after 12 weeks of supplementation.
  Muscle strength was assessed using a handgrip dynamometer to evaluate functional improvement following 12 weeks of supplementation.

SECONDARY OUTCOMES:
Change in Body Weight | Baseline and after 12 weeks of supplementation
  Body weight (kg) was measured using a calibrated digital scale to assess changes in body mass after supplementation.
Change in Body Mass Index | Baseline and after 12 weeks of supplementation.
  BMI (kg/m²) was calculated as weight divided by height squared to evaluate body composition changes.
Change in Serum Globulin Levels | Baseline and after 12 weeks of supplementation.
  Serum globulin concentration (g/dL) was determined using standard biochemical methods to assess protein metabolism changes.

CONTACTS AND LOCATIONS:
Overall Officials: Sérgio H Santos, PhD, Principal Investigator — State University of Minas Gerais
Locations (1):
- State University of Minas Gerais, Montes Claros, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No